CLINICAL TRIAL: NCT01733654
Title: A Multi-center Randomized Double-blind Placebo-controlled Parallel-group Study to Investigate Efficacy and Safety of RO4995819 vs Placebo, as Adjunct Therapy in Patients w/Major Depressive Disorder
Brief Title: Investigate Efficacy & Safety of RO4995819 vs. Placebo as Adjunct Tx in Patients w/Major Depressive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Charles DeBattista, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23708
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Depression; Major Depressive Disorder
Keywords: depression; major depressive disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RO4995819 5mg (Active Comparator): RO4995819 5mgX6wks
  Interventions: Biological: RO4995819
- RO4995819 15mg (Active Comparator): RO4995819 15mg X 6 weeks
  Interventions: Biological: RO4995819
- RO4995819 30mg (Active Comparator): RO4995819 30mg X 6 weeks
  Interventions: Biological: RO4995819
- Placebo (Placebo Comparator): Placebo X 6 weeks
  Interventions: Biological: RO4995819

INTERVENTIONS:
Biological: RO4995819 — The investigation of RO4995819 as adjunctive therapy in MDD patients is supported by preclinical and clinical evidence implicating dysfunction of glutamatergic pathways in the pathophysiology of depression and cognitive disorders, and accumulated evidence of the antidepressant and procognitive effects of mGlu2/3 antagonism.
  Other Names: RO4995819, 5mg; RO4995819, 15mg; RO4995819, 30mg; Placebo, (a pill that does not contain active drug)

SUMMARY:
The purpose of the study is to explore the efficacy of 6 weeks treatment of an investigational medication, RO4995819, versus placebo as adjunctive therapy in patients with major depression.

DETAILED DESCRIPTION:
The investigators hope to learn the efficacy of 6 weeks treatment of RO4995819 versus placebo as adjunctive therapy in patients with MDD having inadequate response to ongoing antidepressant treatment based on mean change in Montgomery Asberg Depression Rating Scale (MADRS) scores from baseline to end of treatment.

This knowledge is valuable because it is a new medication, which may have utility in the population of patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for enrollment in this study if they meet all of the following criteria:

1. An outpatient w/a primary diagnosis of major depressive disorder w/out psychotic features
2. Inadequate response to current, ongoing antidepressant tx of SSRI/SNRI.
3. Having at least 1 but no more than 2 antidepressant treatment failures w/in the index depressive episode
4. Dose/duration of antidepressant treatment in index episode can be verified by documentation from one of following:

   1. Med records;
   2. Pharmacy records;
   3. Treating and/or referring physician (indicating medication, dose, dates of treatment).
5. Documentation of clinical/treatment history must be available.
6. Index depressive episode started w/in 1 year of screening.
7. Confirmed compliance w/current SSRI/SNRI treatment based on blood screen.
8. Existing med regimens should be stable for 6 wks prior to screening
9. 18-65 y.o. at time of consent
10. BMI 18.0 to 35.0 kg/m2 inc.
11. Patients w/reproductive potential must agree to use specified contraceptive protection during tx period and for at least 90 days after last dose of study drug:

    * Males w/partners of childbearing potential or partners must use a barrier method of contraception or remain sexually abstinent.
    * Females who are not either surgically sterile (tubal ligation, removal of ovaries or uterus) or post-menopausal (no spontaneous menstrual periods for at least 1 yr confirmed by a hormone panel [FSH and 17βestradiol])must agree to use 2 adequate methods of contraception, including at least one method w/ failure rate of < 1% per yr (e.g., hormonal implants, combined oral contraceptives, vasectomized partner, abstinence).
12. Able to participate and willing to give written informed consent.

Exclusion Criteria:

Patients are excluded from this study if the answer is 'yes' to any of the following:

Current and past treatment history:

1. Currently receiving tx w/3 or more antidepressants.
2. Currently receiving tx w/prohibited meds.
3. Significant ongoing use of high doses of barbiturates, benzodiazepines or other anxiolytic drugs.
4. Previously received RO4995819.
5. Participated in investigational drug or device study w/in 6 mos of screening or in index depressive episode.
6. History of non-response to Electroconvulsive Therapy (ECT), Vagus Nerve Stimulation (VNS),or Repetitive Transcranial Magnetic Stimulation (RTMS).
7. Planning to begin/change current regimen of individual psychotherapy including cognitive behavioral therapy during the 6 week treatment period of the study and the first 2 weeks of follow-up.
8. Present DSM-IV-TR axis I diagnosis except for anxiety comorbidity
9. Past or present psychotic symptoms.
10. Mood disorder due to medical condition or substance use/abuse/dependence.
11. Established personality disorder
12. Alcohol and/or substance abuse/dependence during the last 6 months.
13. A significant risk for suicidal behavior
14. Past or present neurological disorder.
15. Present eating disorder
16. Abnormal thyroid function.
17. Active upper gastrointestinal tract disease
18. Unstable medical condition that could pose unacceptable risk to the patient in this study.
19. Positive result on hepatitis B (HBV), hepatitis C (HCV), or HIV 1 and 2.
20. Positive test for drugs of abuse.
21. Abnormality on 12-lead electrocardiogram (ECG), including a QTcF of ≥450 milliseconds.
22. Lab abnormality
23. Positive pregnancy test, breast feeding,or intention to become pregnant during the course of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | 6 weeks
  The investigators hope to learn the efficacy of 6 weeks treatment of RO4995819 versus placebo as adjunctive therapy in patients with MDD having inadequate response to ongoing antidepressant treatment based on mean change in Montgomery Asberg Depression Rating Scale (MADRS) scores from baseline to end of treatment. This knowledge is valuable because it is a new medication, which may have utility in the population of patients with major depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Charles DeBattista, DMH, MD, Principal Investigator — Stanford University Department of Psychiatry